CLINICAL TRIAL: NCT02238353
Title: AZE/FLU Nasal Spray on Symptom Control, Nasal Mediators and Nasal Hyperresponsiveness in Allergic Rhinitis (AR)
Brief Title: AZELASTINE/FLUTICASONE (AZE/FLU) Nasal Spray on Symptom Control, Nasal Mediators and Nasal Hyperresponsiveness in Allergic Rhinitis (AR)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: azelastine/fluticasone AZE/FLU
Record Dates: First submitted 2013-08-22; First posted 2014-09-12 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Allergic Rhinitis; House Dust Mite Allergy
MeSH Terms: conditions — Rhinitis, Allergic; Dust Mite Allergy | interventions — azelastine; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- azelastine + fluticasone (Experimental): azelastine 137 µg + fluticasone 50 µg combined applied twice daily one puff in each nostril duration: 4 weeks
  Interventions: Drug: azelastine + fluticasone
- placebo (Placebo Comparator): twice daily one puff in each nostril duration: 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: azelastine + fluticasone
  Other Names: dymista
  Arms: azelastine + fluticasone
Drug: Placebo
  Arms: placebo

SUMMARY:
Comparative analysis of the efficacy of intranasal MP29-02 (a novel formulation of azelastine and FP) has already been conducted in patients with moderate-to-severe seasonal AR. The combination formulation appeared to be superior in these patients with better symptomatic relief. However, objective analysis of the effect of this treatment on nasal mediators and/or nasal hyperreactivity has not yet been performed and would help in understanding the additional benefit of the combination treatment over monotherapy with nasal corticosteroids.

DETAILED DESCRIPTION:
Comparative analysis of the efficacy of intranasal MP29-02 (a novel formulation of azelastine and FP) has already been conducted in patients with moderate-to-severe seasonal AR. The combination formulation appeared to be superior in these patients with better symptomatic relief. However, objective analysis of the effect of this treatment on nasal mediators and/or nasal hyperreactivity has not yet been performed and would help in understanding the additional benefit of the combination treatment over monotherapy with nasal corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an ARIA-based diagnosis of persistent moderate/severe AR (≥ 2 nasal symptoms suggestive of allergic rhinitis and positive skin prick tests to house dust mite (HDM) (HAL Allergy, Leiden, The Netherlands) at screening. Patients with additional seasonal pollen allergies may be included providing that they are included outside their individual pollen season, and with VAS score for total nasal symptoms of more than 5
2. VAS for TNS of more than 5, and rT5SS of more than 8 at both screening and randomization
3. Age > 18 and < 60 years
4. Eosinophilia of more than 5% in nasal secretions at screening
5. Nasal hyperreactivity (drop of PNIF >20 %) at randomization
6. Possibility to give reliable information and written informed consent

Exclusion Criteria:

1. Any evidence of clinically relevant acute or chronic cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrine, metabolic, mental, neurological, or other disease at screening
2. History of allergic reaction to fluticasone propionate, azelastine hydrochloride or one of the excipients (e.g. benzalkonium chloride, phenylethyl alcohol, microcrystalline cellulose)
3. Patients with a change in vision or with a history of increased ocular pressure, glaucoma and/or cataracts
4. Patients with tuberculosis, any type of untreated infection, or recent surgical operation or injury to the nose or mouth
5. Patients on prolonged use of decongestive nose sprays, suffering from so-called rhinitis medicamentosa
6. Patients using other nasal or oral medication affecting nasal function, like nasal corticosteroids, anticholinergics, cromoglycates, leukotriene antagonists, ACE inhibitors during the study or within the last 14 days before randomization; patients using oral corticosteroids during the last 30 days
7. Patients using cytochrome P450 inhibitors (e.g. ritonavir)
8. Nasal endoscopic evidence of rhinosinusitis with or without nasal polyposis (NP) or structural abnormalities such as clinically relevant septal deviation (septum reaching concha inferior or lateral nasal wall) or septal perforation at screening
9. Patients on immunotherapy (IT) for HDM or with history of IT for HDM
10. Patients with a psychiatric, addictive, or any disorder of which the investigators feel that this may compromise the ability to give truly informed consent for participation in this study or provide reliable information on the questionnaire
11. Patients being enrolled in other clinical trials within the last 3 months
12. Pregnancy or breastfeeding
13. Malignancies or severe comorbidity
14. Smoking
15. Use of anticoagulation medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
change in expression of inflammatory mediators (Histamine / Substance P / IL-5 / EPO) | 4 weeks after treatment
  Change in expression of inflammatory mediators (Histamine / Substance P / interleukin 5 (IL-5) / EPO) at after 4 weeks of therapy with AZE/FP or placebo nasal spray.
  Unit of measurement: µg/ml

SECONDARY OUTCOMES:
change in PNIF values upon CDA exposure | 4 weeks treatment
  Nasal hyperreactivity (NHR) can be assessed with peak nasal inspiratory flow (PNIF) measurement before and after cold dry air (CDA) provocation.
  1. Peak nasal inspiratory flow (PNIF) Peak nasal inspiratory flow evaluation is a physiologic measure of air flow through both nasal cavities during forced inspiration. The PNIF can be measured using a portable nasal inspiratory ﬂow meter and is expressed in liters per minute.
  2. Cold dry air (CDA) provocation CDA nasal provocation can be performed by delivering compressed dry air through a mask placed over nose and mouth of the patient, while breathing only through the nose. Patients will be exposed during 15 minutes. NHR is defined as a drop in PNIF larger than 20 % from baseline upon CDA challenge.
  The efficacy of MP29-02 treatment will be evaluated by measuring the change in PNIF values upon CDA exposure in both treatment arms.
  Unit of measurement of PNIF: L/min

OTHER OUTCOMES:
change in assessment of visual analogue scale (VAS) for total nasal symptom (TNS) and individual nasal symptoms, reflective total of 5 symptom scores (rT5SS) and Allergic Rhinitis Control Test (ARCT) | 1 week after treatment
  A Visual Analogue Scale (VAS) is a measurement of patient's subjective evaluation of symptom severity. Patients will score the severity of their total nasal symptoms (TNS) on a scale, as well as each individual nasal symptom (rhinorrhea, pruritis, sneezing, nasal obstruction), with 0 meaning no symptoms and 10 meaning the worst symptoms. The cut off value of 5/10 is to distinguish between controlled and uncontrolled AR.
  Patients will score their reflective nasal and ocular symptoms on a 4-point scale from absent (0), mild (1), moderate (2) to severe (3)). Minimum score: 0/15 as having no trouble with any of the symptoms; and maximum score: 15/15 as having maximum trouble with all the symptoms
  The Allergic Rhinitis Control Test (ARCT): Patients score the five questions from 1 (always troublesome) to 5 (never troublesome). Minimum score: 5/25 ; maximum score: 25/25. A score from 5/25 to 20/25 is assumed not controlled AR; a score higher then 20/25 is assumed controlled.
Effects of therapy with AZE/FP or placebo on nasal inflammatory mediators (Histamine / Substance P (SP) / IL-5 / EPO) | one week after treatment
  Change in expression of inflammatory mediators (Histamine / Substance P / IL-5 / EPO) at after 1 week of therapy with AZE/FP or placebo nasal spray.
  Unit of measurement: µg/ml
change in PNIF values upon CDA exposure | 1 week of treatment
  Nasal hyperreactivity (NHR) can be assessed with peak nasal inspiratory flow (PNIF) measurement before and after cold dry air (CDA) provocation.
  Peak nasal inspiratory flow (PNIF) Peak nasal inspiratory flow evaluation is a physiologic measure of air flow through both nasal cavities during forced inspiration. The PNIF can be measured using a portable nasal inspiratory ﬂow meter and is expressed in liters per minute.
  Cold dry air (CDA) provocation CDA nasal provocation can be performed by delivering compressed dry air through a mask placed over nose and mouth of the patient, while breathing only through the nose. Patients will be exposed during 15 minutes. NHR is defined as a drop in PNIF larger than 20 % from baseline upon CDA challenge.
  The efficacy of MP29-02 treatment will be evaluated by measuring the change in PNIF values upon CDA exposure in both treatment arms.
  Unit of measurement of PNIF: L/min
change in assessment of visual analogue scale (VAS) for total nasal symptom (TNS) and individual nasal symptoms, rT5SS and Allergic Rhinitis Control Test (ARCT) | 4 weeks after treatment
  A Visual Analogue Scale (VAS) is a measurement of patient's subjective evaluation of symptom severity. Patients will score the severity of their total nasal symptoms (TNS) on a scale, as well as each individual nasal symptom (rhinorrhea, pruritis, sneezing, nasal obstruction), with 0 meaning no symptoms and 10 meaning the worst symptoms. The cut off value of 5/10 is to distinguish between controlled and uncontrolled AR.
  Patients will score their reflective nasal and ocular symptoms on a 4-point scale from absent (0), mild (1), moderate (2) to severe (3)). Minimum score: 0/15 as having no trouble with any of the symptoms; and maximum score: 15/15 as having maximum trouble with all the symptoms
  The Allergic Rhinitis Control Test (ARCT): Patients score the five questions from 1 (always troublesome) to 5 (never troublesome). Minimum score: 5/25 ; maximum score: 25/25. A score from 5/25 to 20/25 is assumed not controlled AR; a score higher then 20/25 is assumed controlled.

CONTACTS AND LOCATIONS:
Overall Officials: peter hellings, MD, Principal Investigator — UZ Leuven
Locations (1):
- Uz Leuven Dienst Nko, Leuven, Vlaams Brabant, Belgium